CLINICAL TRIAL: NCT06708897
Title: Phase 1 Study of ZE50-0134 in Relapsed and Refractory Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL), and Select Low-grade Lymphomas
Brief Title: A Phase 1 Study of ZE50-0134 in Relapsed and Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, and Select Low-grad Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lomond Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZE50-0134-0002
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: CLL / SLL; CLL (Chronic Lymphocytic Leukemia); SLL (Small Lymphocytic Lymphoma)
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: dose escalation and dose optimization study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- ZE50-0134 Dose Level -1 (Experimental): Optional and would only be performed Dose Level 1 is poorly tolerated
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Dose Level 1 (Experimental)
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Dose Level 2 (Experimental)
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Dose Level 3 (Experimental)
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Dose Level 4 (Experimental)
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Dose Level 5 (Experimental)
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Selected dose 1 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study
  Interventions: Drug: ZE 50-0134
- ZE50-0134 Selected dose 2 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study
  Interventions: Drug: ZE 50-0134

INTERVENTIONS:
Drug: ZE 50-0134 — oral capsules QD

SUMMARY:
This is a clinical study aiming to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ZE50-0134 in relapsed and refractory chronic lymphocytic leukemia, small lymphocytic lymphoma, and select low-grad lymphomas.

DETAILED DESCRIPTION:
A Phase 1, Open-label, Dose Escalation and Dose Expansion, Multicenter Clinical Trial to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ZE50-0134 in Relapsed and Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, and Select Low-grad Lymphomas. The study is an open-label, with 2 parts.

Part 1 will utilize a 3+3 design. Eligible patients will be sequentially enrolled into each of 5 planned dose level cohorts. The purpose of Part 1 dose escalation is to determine the maximum tolerated dose of ZE50-0134.

IPart 2 is a dose expansion of ZE50-0134 and will include two distinct doses who are venetoclax naïve treated at either the Biologically Effective Dose or Maximum Tolerated Dose and one dose lower. The purpose of Part 2 is to determine the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary antitumor activity of ZE50-0134 in subjects with CLL/SLL.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years.
2. Disease as defined below:

   Part 1: Patients with symptomatic CLL or SLL (defined by iwCLL) without del(17p)/TP53 must have received ≥2 prior therapies that have included a BTKi and venetoclax (or declined this) or Patients with progressive low-grade lymphoma that includes marginal zone lymphoma, lymphoplasmacytic lymphoma (including Waldenstrom's macroglobulinemia) who have received at least 2 therapies including a BTKi and CD20 antibody-based therapy.

   Part 2: Patients with symptomatic CLL or SLL (defined by iwCLL) must have received ≥1 prior therapies that have included a BTKi and be venetoclax naive.
3. Prior to beginning part 2, an activation amendment will be submitted to the FDA that includes safety, pharmacokinetics, pharmacodynamics and early efficacy data from the Part 1 portion. At this time, we may also include cohorts of specific types of low-grade lymphoma as well. Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements to be conducted within 7 days before the first dose of study drug:

   * Absolute neutrophil count (ANC) > 0.75 x 109/L. For subjects with documented bone marrow involvement ≥ 0.5 x 109/L
   * Platelet count > 50 x 109/L. For subjects with documented bone marrow involvement ≥ 30 x 109/L
   * Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 x ULN
   * Creatinine or Cystatin C glomerular filtration rate (GFR) ≥60 mL/min. Estimated GFR (eGFR) according to the Modification of Diet in Renal Disease Study Group (MDRD) formula and expressed in mL/min. To convert mL/min/1.73 m2 to mL/min multiply by the individual's BSA calculated using an appropriate formula and divide by 1.73 Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less Negative serum or urine pregnancy test must be obtained within 7 days before the first dose of study drug in women of childbearing potential. Negative results must also be available before each cycle.

Postmenopausal women, as defined below, are exempt from pregnancy testing:

* Age >50 years with amenorrhea for at least 12 months or
* Age ≤50 years with 6 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within postmenopausal range (>40 mIU/mL) OR
* Permanently sterilized women (e.g., hysterectomy, bilateral salpingectomy, or uterine ablation) Women and men of reproductive potential must agree to use highly effective contraception when sexually active. This applies for the period between signing of the informed consent and 90 days after the last administration of study drug. These methods should be documented in source documents. The investigator or a designated associate is requested to advise the subject on how to achieve highly effective birth control. Ability to understand and the willingness to sign a written informed consent. A signed informed consent (including consent for genetic biomarker

Exclusion Criteria:

Subjects will be excluded from the study if they display any of the following criteria:

1. FOR PART 2 ONLY

   - No prior venetoclax treatment

   FOR BOTH PARTS ALL THE FOLLOWING APPLY:
2. Know active Richter's transformation. Patients who have been treated for this diagnosis and have been in remission for > 2 years without evidence of this and who have only CLL are considered eligible
3. Known hypersensitivity to the study drug or excipients of the preparation or any agent given in association with this study.
4. Clinically significant cardiac disease including congestive heart failure > New York Heart Association (NYHA) Class II, evidence for uncontrolled coronary artery disease (e.g., unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months or myocardial infarction within the past 6 months before first dose, major regional wall motion abnormalities upon baseline echocardiography), and cardiac arrhythmias requiring anti- arrhythmic therapy except for beta-blockers and digoxin.
5. Known Active cytomegalovirus (CMV), hepatitis B or C virus infection.
6. Known Active SARS-CoV-2 infection; prior SARS-CoV-2 infection allowed if completely recovered > 14 days.
7. Active clinically serious infections of Grade >2, requiring parenteral therapy; Subjects may be eligible after infection resolves.
8. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura within 28 days of enrolment.
9. Allogeneic bone marrow transplant within 4 months before first dose of study drug (Subjects must have completed immunosuppressive therapy before enrollment).
10. Active cancer that limits expected survival to < 2 years or requires active therapy concomitant with this treatment. Exclusions would be localized skin cancer, breast cancer, prostate cancer that are resected or malignancies treated with hormonal or immune therapies alone. All cases of secondary cancer should be discussed with the medical monitor.
11. A physical exam or laboratory finding that contraindicates the use of investigational therapy or otherwise places the subject at excessively high risk for treatment, as determined by the investigator. A discussion between the investigator and sponsor regarding eligibility is encouraged for such cases.
12. Unresolved toxicity of previous treatments (excluding cases of alopecia) Grade ≥2.
13. Requires ongoing immunosuppressive therapy, including systemic (e.g., intravenous or oral) corticosteroids for the treatment of cancer or other conditions. Note: Subjects may use topical or inhaled corticosteroids or low-dose steroids (≤10 mg of prednisone or equivalent per day) as therapy for comorbid conditions. Short courses of steroids before first dose are allowed for tumor flare.
14. Major surgery or significant trauma within 4 weeks before the first dose of study drug.
15. Breastfeeding women: breastfeeding women have to discontinue breastfeeding before onset of and during treatment and should be discontinued for at least 3 months after end of treatment.
16. Subjects with QTcF > 470 msec that cannot be corrected with electrolyte replacement, hydration, or medication modifications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | Up to 24 cycles, 4 weeks each
  Frequency, severity, and relationship to study drug of any TEAEs or abnormalities of laboratory tests; SAEs; and AEs leading to discontinuation of study treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 cycles, 4 weeks each
  The ORR is defined as the proportion of subjects who have a best overall response of PR or better as determined by investigators using the iwCLL guidelines, Lugano guidelines, or Waldenstrom guidelines.
Assess duration of response (DOR) | Up to 24 cycles, 4 weeks each
  DOR is defined in responders as the time from documentation of tumor response (date of first PR or better response) to the date of disease progression as determined by the investigator using iwCLL guidelines, Lugano guidelines, Waldenstrom guidelines or death due to any cause.
Progression-free survival (PFS) | Up to 24 cycles, 4 weeks each
  PFS is defined as time from first dose until progression as assessed by the investigator using iwCLL guidelines, Lugano guidelines or death due to any cause.
Time to next treatment (TTNT) | Up to 24 cycles, 4 weeks each
  TTNT is defined as time from first dose to the initiation of alternative treatment other than ZE50-0134 for CLL or death.
ZE50-0134 blood plasma concentration | 2 cycles, 4 weeks each
  ZE50-0134 blood plasma concentration

OTHER OUTCOMES:
Caspase 3 activation level | 3 cycles, 4 weeks each
  Measuring caspase 3 activation in CLL and lymphoma cells
Immune cells count | 3 cycles, 4 weeks each
  Serial immune CD8 T-cells, NK cells, and normal B-cells during ZE50-0134 therapy
Rate of undetectable Measurable residual disease (uMRD) response in bone marrow and blood | 12 cycles, 4 weeks each
  Rate of uMRD is defined as the proportion of evaluable subjects with MRD undetectable in bone marrow and blood

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio